CLINICAL TRIAL: NCT01883921
Title: Gamma Globulin Observations and Outcomes Database for Specific Home Infusion Evidence, Patient Care And Research Data in Patients With Primary Immunodeficiency Disease (GOOD-SHEPARD-PI)
Brief Title: Gamma Globulin Observations and Outcomes Database for Patients With Primary Immunodeficiency Disease (GOOD-SHEPARD-PI)
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: BriovaRx Infusion Services (Industry)
Responsible Party: Principal Investigator, Timothy P. Walton, MHS, CCRP, Timothy P. Walton, MHS, CCRP, BriovaRx Infusion Services
Other Study IDs: BIS1-13-002
Record Dates: First submitted 2013-06-19; First posted 2013-06-21 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: Primary Immunodeficiency; Immunodeficiencies; Primary Immunodeficiency Diseases; PIDD; CVID; PI; Common Variable Immunodeficiency; Hypogammaglobulinemia; Acquired Hypogammaglobulinemia; Immunology; Autoimmune Deficiency; Intravenous Immunoglobulin; Subcutaneous Immunoglobulin; IVIg; SCIg; Immune Globulin; Outcomes Research; Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immunologic Deficiency Syndromes; Common Variable Immunodeficiency; Agammaglobulinemia | interventions — Immunization, Passive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunoglobulin Therapy
  Interventions: Other: Immunoglobulin Therapy

INTERVENTIONS:
Other: Immunoglobulin Therapy

SUMMARY:
Primary:

* Demonstrate the utility of an electronic data capture (EDC) system (CareExchange™) using infusion nurse and patient measured physical, quality of life (QOL), respiratory, laboratory, and disability assessments in patients with Primary Immunodeficiency Disease (PIDD).

Secondary:

* Change in Intravenous/Subcutaneous Immunoglobulin (IVIg/SCIg) dose effects measured outcomes.
* Change in IVIg/SCIg dose timing effects measured outcomes.
* Change in patient status is reflected in measured outcomes.
* Assess the value to physicians from collected outcomes data.
* Identify types of patients by response to IVIg/SCIg therapies (well maintained, problematic, etc.).
* Change in response rate as measured by outcomes to IVIg/SCIg therapies by disease state, co-morbidities, and demographics.

DETAILED DESCRIPTION:
This is a prospective, observational evaluation of immunoglobulin (Ig) therapy in consenting PIDD adult and assenting pediatric subjects who receive infusion services from BriovaRx Infusion Services (formerly AxelaCare Health Solutions, LLC). Subjects meeting all inclusion criteria who have provided informed consent/assent for trial participation will have validated, physician-prescribed, standard-of-care outcome measures, and Ig administration information recorded during normal home infusion visits. There will also be standard-of-care questions captured within some outcome measures recorded during normal home infusion visits that may be at a frequency and/or combination which may not be considered routine clinical care by some physicians who treat for this medical condition. Collected data will be de-identified and aggregated into cohorts of like diagnosis for trend analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any form of Primary Immunodeficiency Disease
* Age at enrollment ≥ 7
* Sign informed consent/assented to participation
* Ability to read and write English
* Understanding of study procedures and ability to comply with study procedures for the entire length of the study
* Receiving Ig under the discretion of the patient's treating physician in accordance with standard treatment practices
* Have been on or is between doses of Ig under the discretion of the patient's treating physician in accordance with standard treatment practices
* Being considered to be prescribed Ig under the discretion of the patient's treating physician in accordance with standard treatment practices
* Determined to be eligible for infusion services by BriovaRx Infusion Services (formerly AxelaCare Health Solutions, LLC.) in collaboration with the patient's prescribing physician

Exclusion Criteria:

* Children (age ≤ 6 years)
* Prisoners, and other wards of the state
* Determined to have non-competency of data collection requirements (physical assessments and use of an iPAD™) by the study participant's caregiver

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who is aged 7 years or greater at time of enrollment; who is on Ig therapy, have been on or is between doses of Ig therapy, or is being considered to be prescribed Ig therapy; provides informed consent for participation; and who has been determined to be eligible for infusion services by BriovaRx Infusion Services (formerly AxelaCare Health Solutions, LLC), in collaboration with the patient's prescribing physician. Subjects will be recruited from the practices of participating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Analysis of collected data captured in CareExchange™ -ability to show and track changes in outcome data in PIDD patients. | Up to 5 Years

SECONDARY OUTCOMES:
Physician feedback will demonstrate if having real-time access to patient data captured during a home infusion will assist in the management of the patient's disease. | Up to 5 Years
Response rate for those receiving IVIg/SCIg therapies. | Up to 5 Years
Exhibit differences in response rate of IVIg/SCIg therapies across disease states and demographics | Up to 5 Years
Measure variables within patients who receive IVIg/SCIg therapies | Up to 5 Years

CONTACTS AND LOCATIONS:
Locations (1):
- BriovaRx Infusion Services, Lenexa, Kansas, United States